CLINICAL TRIAL: NCT07262255
Title: WATCHMAN FLX Pro European Registry
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Boston Scientific Corporation (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Prevention
Other Study IDs: S2603
Record Dates: First submitted 2025-11-17; First posted 2025-12-03 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Non-valvular Atrial Fibrillation (AF); Left Atrial Appendage Closure
Keywords: LAAC
MeSH Terms: interventions — Left Atrial Appendage Closure

STUDY DESIGN:
Intervention Model Description: Registry
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- WATCHMAN FLX Pro (Other): This arm is intended to gather real world clinical data for patients undergoing left atrial appendage closure (LAAC) with the WATCHMAN FLX™ Pro device.
  Approximately 300 patients undergo the LAAC procedure in conjunction with the use of the VersaCross Connect™ LAAC Access Solution.
  Interventions: Device: Left atrial appendage closure

INTERVENTIONS:
Device: Left atrial appendage closure — The WATCHMAN FLX Pro LAAC Technology is intended to prevent thrombus embolization from the left atrial appendage and reduce the risk of life-threatening bleeding events in adult patients with non-valvular atrial fibrillation who are eligible for anticoagulation therapy or who have a contraindication to anticoagulation therapy.
  The VersaCross Connect™ LAAC Access Solution is indicated for the percutaneous introduction of various types of cardiovascular catheters and guidewires to all heart chambers, including the left atrium via transseptal perforation / puncture.

SUMMARY:
The WATCHMAN FLX Pro European registry is intended to gather real world clinical data for patients undergoing left atrial appendage closure (LAAC) with the WATCHMAN FLX™ Pro device. In a subregistry with approximately 300 patients, it is intended to use the VersaCross Connect™ LAAC Access Solution.

ELIGIBILITY:
Inclusion Criteria:

1. Subject is attempted to be treated with the WATCHMAN FLX™ Pro LAAC device.
2. Subject has non-valvular atrial fibrillation (i.e., atrial fibrillation in the absence of moderate or greater mitral stenosis or a mechanical heart valve) and is clinically indicated for a WATCHMAN FLX™ Pro LAAC device, per the Instructions for Use (IFU).
3. Subject or legal representative who are willing and capable of providing informed consent.
4. Subject is able and willing to return for required follow-up visits and examinations.
5. Subject whose age is 18 years or above, or who is of legal age to give informed consent specific to state and national law.

Exclusion Criteria:

1. Subject has a documented life expectancy of less than 12 months.
2. Subject who is currently enrolled in another investigational study or registry except when the subject is participating in a mandatory governmental registry, or a purely observational registry with no associated treatments.
3. Intracardiac thrombus is present.
4. An atrial septal defect repair or closure device or a patent foramen ovale repair or closure device is present.
5. The LAA anatomy will not accommodate a Closure Device.
6. Subject has a known hypersensitivity or contraindications according to IFU.
7. Subject is of childbearing potential and is, or plans to become, pregnant during the time of the study.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2025-12-17 (Actual); Primary Completion 2027-08 (Estimated); Study Completion 2028-09 (Estimated)

PRIMARY OUTCOMES:
Number of participants with a safety event treated with the WATCHMAN FLX Pro | Between the time of procedure and within 7 days following the procedure or by hospital discharge, whichever is later
  Proportion of subjects with one or more of the following events between the time of procedure and within 7 days following the procedure or by hospital discharge, whichever is later: all-cause death, ischemic stroke, systemic embolism, or device or procedure related events requiring open cardiac surgery or major endovascular intervention such as pseudoaneurysm repair, AV fistula repair, or other major endovascular repair.
  Percutaneous catheter drainage of pericardial effusions, snaring of an embolized device, thrombin injection to treat femoral pseudoaneurysm and minor nonsurgical treatments of access site complications are excluded from this endpoint.
Number of participants with a safety event treated with the VersaCross Connect™ LAAC Access Solution | Between the time of procedure and within 7 days following the procedure or by hospital discharge, whichever is later
  Proportion of subjects with one or more of the following events between the time of procedure and within 7 days following the procedure or by hospital discharge, whichever is later:
  For all enrolled subjects, who had an attempt to insert the VersaCross Connect™ LAAC Access Solution device, the composite rate of all-cause death, all stroke, systemic embolism, pericardial effusion resulting in interventions*, and ISTH major bleeding.
  *Pericardial effusion/tamponade requiring pericardiocentesis or surgery to treat
Number of participants with a successful VersaCross Connect™ LAAC Access Solution treatment | Completion of transseptal puncture
  VersaCross Connect™ LAAC Access Solution acute procedural success: Acute Procedural Success is defined as transseptal puncture success (VersaCross RF-wire crossing into left atrium).

CONTACTS AND LOCATIONS:
Overall Officials: Marek Grygier, Prof. MD, PHD, Principal Investigator — Uniwersytecki Szpital Kliniczny w Poznaniu; Arian Sultan, Prof. MD, Principal Investigator — Asklepios Klinik Saint Georg
Locations (2):
- Spain (2):
  - Hospital de Leon, León
  - Clinica Universidad de Navarra, Pamplona

IPD SHARING:
Plan to Share IPD: No